CLINICAL TRIAL: NCT01781793
Title: Mechanisms of Exertional Dyspnea in Fibrotic Interstitial Lung Disease
Acronym: Dyspnea_ILD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: H13-00059
Record Dates: First submitted 2013-01-28; First posted 2013-02-01 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Lung; Disease, Interstitial, With Fibrosis
Keywords: dyspnea, exercise endurance, lung disease
MeSH Terms: conditions — Disease; Dyspnea; Lung Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fibrotic ILD Patients, Room Air (Placebo Comparator): Fibrotic ILD patients will breathe room air (21% oxygen) during a constant work rate exercise test
  Interventions: Other: Room air
- Fibrotic ILD Patients, Hyperoxia (Active Comparator): Fibrotic ILD patients will breathe hyperoxia (60% oxygen) during a constant work rate exercise test
  Interventions: Other: Hyperoxia

INTERVENTIONS:
Other: Room air — Humidified room air (21% oxygen) will be inspired
  Arms: Fibrotic ILD Patients, Room Air
Other: Hyperoxia — 60% oxygen will be inspired
  Arms: Fibrotic ILD Patients, Hyperoxia

SUMMARY:
Exertional dyspnea is a major source of crippling distress and is the hallmark symptom of fibrotic interstitial lung disease (ILD). Due to the scientific community's poor understanding of the pathophysiological mechanisms of dyspnea there are no therapeutic interventions that consistently reduce dyspnea in this population. The investigators aim to determine the physiological mechanisms of exertional dyspnea in patients with fibrotic ILD and the impact of hyperoxia on exertional dyspnea and exercise endurance. This study will likely identify an important physiological mechanism of dyspnea in fibrotic ILD and may contribute to the development of effective therapies to reduce dyspnea in this population.

The central hypothesis is that dyspnea in fibrotic ILD is primarily a result of an imbalance between the drive to breathe and the tidal volume response of the respiratory system (i.e., neuromechanical uncoupling) and that experimental reduction of neuromechanical uncoupling via hyperoxic breathing will reduce exertional dyspnea and improve exercise endurance.

DETAILED DESCRIPTION:
The purpose of this study is to determine the physiological mechanisms of shortness of breath (dyspnea) in patients with fibrotic Interstitial Lung Disease (ILD) and to determine how breathing supplemental oxygen can manipulate these mechanisms to improve dyspnea and exercise capacity.

The research question is twofold: (Aim 1) To determine the physiological mechanisms of exertional dyspnea in patients with fibrotic ILD; (Aim 2) To determine the effects of hyperoxia on exertional dyspnea and exercise endurance in patients with fibrotic ILD.

Experimental Overview: Participants with fibrotic ILD and control participants will report to the exercise laboratory on four separate occasions separated by a minimum of 48 hours between visits. On visit 1, participants and control participants will complete medical history screening, chronic activity-related dyspnea questionnaires, anthropometric measurements, pulmonary function assessment, and a symptom limited incremental cycle exercise test for familiarization purposes. On visit 2, participants and control participants will perform pulmonary function testing followed by another incremental cycle exercise test. Detailed physiological and sensory measurements will be obtained on both visits but the primary analysis will be based on visit 2 results. Data from visit 2 will address the Aim 1. Visits 3 and 4 will include pulmonary function testing followed by a constant-load cycle exercise test at 75% of peak incremental work rate while breathing, in randomized order, either room air or hyperoxia (60% oxygen). Participants and control participants breathing hyperoxia on visit 3 will breathe room air on visit 4 and vice versa while being blinded to the gas concentration. A multi-pair electrode catheter that combines two balloons will be inserted into the esophagus and near infrared spectroscopy will be used to measure tissue oxygenation on visits 2, 3 and 4. Data from visits 3 and 4 will address Aim 2.

Measurements:

* Pulmonary Function: simple spirometry, plethysmography, diffusing capacity, maximum respiratory pressures, static compliance and recoil pressure will be performed on visit 1. Pulmonary function testing on visits 2-4 will only include spirometry and plethysmography so that total lung capacity and vital capacity can be obtained for the determination of operating lung volumes.
* Dyspnea Evaluation: Dyspnea intensity and perceived leg discomfort will be evaluated at rest, every minute during exercise, and at peak exercise using the modified 10-point Borg scale on all testing visits. Upon exercise cessation, subjects will be asked to verbalize their main reason(s) for stopping exercise (i.e., breathing discomfort, leg discomfort, combination of breathing and legs, or some other reason) and to select qualitative descriptors of breathlessness using an established questionnaire.
* Cardio-respiratory Responses to Exercise: Standard cardio-respiratory measures, including minute ventilation, oxygen consumption (VO2), carbon dioxide production, partial pressure of end-tidal carbon dioxide, tidal volume (VT), and breathing frequency.
* Operating volumes will be derived from dynamic inspiratory capacity (IC) manoeuvres. Arterial oxygen saturation will be measured using pulse oximetry. Electrocardiography and blood pressure will be monitored for safety purposes.
* Respiratory Mechanics: Diaphragmatic electromyography (EMGdi) will be measured using a multi-pair electrode catheter that combines two balloons for measuring esophageal and gastric pressures. The ratio of EMGdi to EMGdimax will be used as an index of neural respiratory drive. The ratio between VT and vital capacity (VC) will be used to represent the mechanical response of the respiratory system. Normalizing for EMGdimax and VC allows the stimulus intensity to be standardized and compared across individuals. Thus neuromechanical uncoupling of the respiratory system will be determined as the ratio (or interaction) between neural drive and the mechanical response of the respiratory system (EMGdi/EMGdimax : VT/VC).
* The mechanical work of breathing (WOB) will be calculated as the area within ensemble averaged esophageal pressure-volume loops.

Statistical Analysis:

Aim 1: Exercise-response slopes (e.g., Borg/VO2) will be determined. Briefly, the investigators will obtain the slope from a plot of Borg vs. VO2 for each participant's and control participant's incremental exercise test performed on visit 2. The investigators will determine the bivariate association of Borg/VO2 slope with VO2 slopes of neuromechanical uncoupling, drive to breathe, and VT response using Spearman correlation coefficients. The investigators will then force all three predictor variables into a multivariate linear regression model with Borg/VO2 slope as the outcome variable in order to identify the independent association of neuromechanical uncoupling with exertional dyspnea. Variables will be transformed to approximate a normal distribution if necessary and predictor variables reaching statistical significance will be assessed for a linear relationship with the outcome variable.

Aim 2: The investigators will first use a paired t-test to identify changes in dyspnea and exercise time comparing room air breathing to hyperoxia during constant-load exercise tests on visits 3 and 4. Multivariate models will then be developed using the between-test difference in Borg dyspnea scale and exercise time for each individual as the outcome variables. Predictor variables will include the between-test difference in neuromechanical uncoupling and its individual components. Outcome and predictor variables for the dyspnea outcome will be based on the between-test difference of these variables at iso-time (i.e., the maximum time for which the patient exercised for both the room air and hyperoxia tests). Predictor variables for exercise time will be measured at the end of the test.

As exploratory analyses, the investigators will repeat the above multivariate linear regression analyses in the IPF subgroup, and the investigators will add a categorical ILD subgroup variable to these analyses in order to identify other inter-group differences. Additional adjustment for potential confounders (e.g., sex, body mass index, high resolution computed tomography fibrosis score) will be used in these exploratory analyses if the subgroup sample size is sufficient. A p value < 0.05 will be considered significant for all analyses. Data analysis will be performed using Stata v11.2 (StataCorp, Texas, USA).

ELIGIBILITY:
Inclusion Criteria - Fibrotic ILD participants:

* A multidisciplinary diagnosis of idiopathic pulmonary fibrosis (IPF), idiopathic fibrotic non-specific interstitial pneumonia (NSIP), chronic hypersensitivity pneumonitis (HP), or unclassifiable interstitial lung disease (ILD) with a differential diagnosis that consists of the above diagnoses
* Fibrosis on high resolution computed tomography (HRCT): honeycombing, reticulation, or traction bronchiectasis
* Oxygen saturation ≥ 92% by pulse oximetry at rest while breathing room air

Exclusion Criteria - Fibrotic ILD Participants:

* Concurrent participation in or recent completion (less than 6 weeks) of pulmonary rehabilitation
* A significant lung disease other than fibrotic ILD that, based on clinical assessment, could impair your ability to exercise
* Significant emphysema
* Pulmonary hypertension (high blood pressure in your lungs' arteries)
* Prednisone (a corticosteroid medication) in excess of 10mg/day for at least two weeks within three months of the first study visit
* An ulcer or tumor in your esophagus, or a nasal septum deviation
* Had recent nasopharyngeal surgery
* A cardiac pacemaker
* Allergies to latex and sensitivities to local anaesthetics
* Current smokers or smoked more than 20 packs per year in the past

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
To determine the physiological mechanisms of exertional dyspnea (Aim 1) and the effects of hyperoxia on dyspnea and cycle endurance in patients with fibrotic ILD (Aim 2) | Parameters will be measured during the four visits. Each visit is separated by at least 48 hours and all visits will be completed within 8 weeks. During the course of each visit, parameters will be measured at rest and during the exercise intervention.
  Included will be 16 patients with fibrotic ILD who have no other pulmonary or extra-pulmonary limitation to exercise. Patients will perform an incremental symptom-limited cardio-pulmonary exercise test while detailed ventilatory, metabolic, respiratory mechanical, neuromechanical and sensory responses are measured. Patients will perform a cross-over study with two symptom-limited constant-load cycle exercise tests on separate days at 75% of peak incremental work rate. These tests will be performed breathing room air on one visit and hyperoxia on the other. Detailed physiological and sensory responses will be measured. Multivariate linear regression will be used to identify the association between neuromechanical uncoupling and exertional dyspnea, adjusting for the individual components of neuromechanical uncoupling (i.e., drive to breathe and tidal volume response) (Aim 1). Paired t-tests will be used to compare outcomes between room air and hyperoxic tests (Aim 2).

SECONDARY OUTCOMES:
To determine the mechanism by which hyperoxia improves exertional dyspnea and exercise time | Parameters will be measured during the four visits. Each visit is separated by at least 48 hours and all visits will be completed within 8 weeks. During the course of each visit, parameters will be measured at rest and during the exercise intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan A Guenette, PhD, Principal Investigator — UBC James Hogg Research Centre
Locations (1):
- UBC James Hogg Research Centre, St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Schaeffer MR, Ryerson CJ, Ramsook AH, Molgat-Seon Y, Wilkie SS, Dhillon SS, Mitchell RA, Sheel AW, Khalil N, Camp PG, Guenette JA. Effects of hyperoxia on dyspnoea and exercise endurance in fibrotic interstitial lung disease. Eur Respir J. 2017 May 25;49(5):1602494. doi: 10.1183/13993003.02494-2016. Print 2017 May. No abstract available. PMID 28546272